CLINICAL TRIAL: NCT05945017
Title: Probiotics and the Neurodevelopment in the Premature Infant <32 Weeks Gestational Age and <1500g
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Collaborators: Hospital Clinic of Barcelona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HCB/2021/0454
Record Dates: First submitted 2023-05-19; First posted 2023-07-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Infant, Newborn, Diseases; Infant Development
Keywords: Probiotics; Bifidobacterium bifidum; Lactobacillus acidophilus; Neurodevelopment; Prematurity; Late-onset sepsis
MeSH Terms: conditions — Infant, Newborn, Diseases; Premature Birth

STUDY DESIGN:
Intervention Model Description: Sequential study with consecutive recruitment with a washout period of 12 months between groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bifidobacterium bifidum NCDO 2203 and Lactobacillus acidophilus NCDO 1748 (Experimental): Daily dose of 6x109 UFC Infloran® -Berne, Switzerland- (Bifidobacterium bifidum NCDO 2203 and Lactobacillus acidophilus NCDO 1748) from 7 days of life until reaching a postmenstrual age of 34 weeks or discharge
  Interventions: Dietary Supplement: Infloran® -Berne, Switzerland- (Bifidobacterium bifidum NCDO 2203 and Lactobacillus acidophilus NCDO 1748
- Control (No Intervention): Untreated control group

INTERVENTIONS:
Dietary Supplement: Infloran® -Berne, Switzerland- (Bifidobacterium bifidum NCDO 2203 and Lactobacillus acidophilus NCDO 1748
  Arms: Bifidobacterium bifidum NCDO 2203 and Lactobacillus acidophilus NCDO 1748

SUMMARY:
Unicentric, quasi-experimental, cohort study to evaluate the effect of combining two probiotics (Bifidobacterium bifidum NCDO 2203 and Lactobacillus acidophilus NCDO 1748) in the neurodevelopment of preterm neonates below 32 weeks' gestation and a birthweight under 1,500 g. This probiotic combination has shown to be safe and beneficial in premature neonates in the prevention of NEC. The investigators hypothesised that this mixture would contribute to better neurodevelopmental outcomes of preterm neonates when assessed at 24 months corrected age. Additionally, neurodevelopment improved would be more relevant at 6 years of age, together with a better pattern of neuronal plasticity biomarkers.

Secondarily, this mixture of probiotics could reduce NEC, LOS, intraventricular haemorrhage and neonatal mortality in accordance with previous studies.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants under 32 weeks gestational age and less than 1500g birthweight.
* Born at BCNatal Hospital Clínic between years 2014-2019.

Exclusion Criteria:

* All neonates presenting with suspected congenital anomalies, inborn errors of metabolism, or genetic defects were excluded.
* Infants with a suspected syndrome, or who have suffered events beyond the neonatal period, not related to prematurity, that could entail impairment in neurodevelopment (severe cranioencephalic trauma, oncological process, meningitis, or exposure to toxic substances)

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 233 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Degree of neurodevelopment at 24 months corrected age | 24 months
  Normal neurodevelopment will be considered when no muscle tone changes, no impaired fine or gross motor coordination, Bayley scale score between above 84, no behaviour disorders or visual disability.
Degree of neurodevelopment at 24 months corrected age | 24 months
  Mild impairment will be considered if any of the following: muscle tone changes, impaired fine or gross motor coordination, Bayley scale score between 71-84, moderate behaviour disorders or mild visual disability.
Degree of neurodevelopment at 24 months corrected age | 24 months
  Moderate impairment will be diagnosed when suffering from any of the following: spastic diplegia, hemiplegia, seizures (non-febrile), Bayley scores between 50-70, severe behaviour disorders, moderate visual disability or mild-moderate hypoacusis.
Degree of neurodevelopment at 24 months corrected age | 24 months
  Severe impairment will be attributed to subjects with any of the following: spastic quadriplegia, choreoathetosis, ataxia, Bayley score <50, blindness or severe hypoacusis
Degree of neurodevelopment at 6 years of age | 6 years
  Wechsler Intelligence Scale for Children - Fifth edition. Ranges from below 69 to above 130. Scores from 90-109 indicate average, above it indicates above average and below, below average performance.
Degree of neurodevelopment at 6 years of age | 6 years
  Child behaviour checklist 6-18 years of age. 113 items about behaviour and social competence scored from 0 "absent" to 2 "occurs often"
Degree of neurodevelopment at 6 years of age | 6 years
  Behavior Rating Inventory of Executive Function, Second Edition (BRIEF2). Parent/teacher self reporting form.
Neuroplasticity biomarkers and intestinal permeability | 6 years
  NeuN, Doublecortin, GFAP, GDNF, Ki67, Nrf2, BDNF, NGF, neurotrophin-1 (NT-1), neurotrophin-3 (NT-3), neurotrophin-4 (NT-4), DYRK1A, HIF1α, S100B i GSK3B. IL1B, IL6, IL8, IL10, IL12, TNF- α

SECONDARY OUTCOMES:
Incidence of necrotising enterocolitis | 40 weeks
  cases fulfilling the stage II or above of the modified Bell's Criteria
Mortality | 40 weeks
  Proportion of dead participants before discharge
Incidence of late onset sepsis | 40 weeks
  positive blood culture beyond 72 hours of life
Incidence of Intraventricular haemorrhage | 40 weeks
  Grade I-IV
Intensive care length of stay | 40 weeks
  Days of intensive care

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin James Baucells, MD, Principal Investigator — Neonataology Service, BCNatal Hospital Clínic; Giorgia Sebastiani, Principal Investigator — Neonatology Service, BCNatal Hospital Clínic
Locations (1):
- Neonataology Service, BCNatal Hospital Clinic Seu Maternitat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sjogren YM, Jenmalm MC, Bottcher MF, Bjorksten B, Sverremark-Ekstrom E. Altered early infant gut microbiota in children developing allergy up to 5 years of age. Clin Exp Allergy. 2009 Apr;39(4):518-26. doi: 10.1111/j.1365-2222.2008.03156.x. Epub 2009 Feb 9. PMID 19220322
- [Background] O'Reilly H, Johnson S, Ni Y, Wolke D, Marlow N. Neuropsychological Outcomes at 19 Years of Age Following Extremely Preterm Birth. Pediatrics. 2020 Feb;145(2):e20192087. doi: 10.1542/peds.2019-2087. Epub 2020 Jan 10. PMID 31924688
- [Result] Food and Agricultural Organization of the United Nations and World Health Organization. Health and nutritional properties of probiotics in food including powder milk with live lactic acid bacteria. World Health Organization, (2001).
- [Result] Navarro-Tapia E, Sebastiani G, Sailer S, Toledano LA, Serra-Delgado M, Garcia-Algar O, Andreu-Fernandez V. Probiotic Supplementation During the Perinatal and Infant Period: Effects on Gut Dysbiosis and Disease. Nutrients. 2020 Jul 27;12(8):2243. doi: 10.3390/nu12082243. PMID 32727119
- [Result] Mai V, Young CM, Ukhanova M, Wang X, Sun Y, Casella G, Theriaque D, Li N, Sharma R, Hudak M, Neu J. Fecal microbiota in premature infants prior to necrotizing enterocolitis. PLoS One. 2011;6(6):e20647. doi: 10.1371/journal.pone.0020647. Epub 2011 Jun 6. PMID 21674011
- [Result] Underwood MA, Sohn K. The Microbiota of the Extremely Preterm Infant. Clin Perinatol. 2017 Jun;44(2):407-427. doi: 10.1016/j.clp.2017.01.005. Epub 2017 Mar 22. PMID 28477669
- [Result] Thomas JP, Raine T, Reddy S, Belteki G. Probiotics for the prevention of necrotising enterocolitis in very low-birth-weight infants: a meta-analysis and systematic review. Acta Paediatr. 2017 Nov;106(11):1729-1741. doi: 10.1111/apa.13902. Epub 2017 Jun 9. PMID 28471478
- [Result] Baucells BJ, Mercadal Hally M, Alvarez Sanchez AT, Figueras Aloy J. [Probiotic associations in the prevention of necrotising enterocolitis and the reduction of late-onset sepsis and neonatal mortality in preterm infants under 1,500g: A systematic review]. An Pediatr (Barc). 2016 Nov;85(5):247-255. doi: 10.1016/j.anpedi.2015.07.038. Epub 2015 Nov 21. Spanish. PMID 26611880
- [Result] Bi LW, Yan BL, Yang QY, Li MM, Cui HL. Which is the best probiotic treatment strategy to prevent the necrotizing enterocolitis in premature infants: A network meta-analysis revealing the efficacy and safety. Medicine (Baltimore). 2019 Oct;98(41):e17521. doi: 10.1097/MD.0000000000017521. PMID 31593123
- [Result] van den Akker CHP, van Goudoever JB, Shamir R, Domellof M, Embleton ND, Hojsak I, Lapillonne A, Mihatsch WA, Berni Canani R, Bronsky J, Campoy C, Fewtrell MS, Fidler Mis N, Guarino A, Hulst JM, Indrio F, Kolacek S, Orel R, Vandenplas Y, Weizman Z, Szajewska H. Probiotics and Preterm Infants: A Position Paper by the European Society for Paediatric Gastroenterology Hepatology and Nutrition Committee on Nutrition and the European Society for Paediatric Gastroenterology Hepatology and Nutrition Working Group for Probiotics and Prebiotics. J Pediatr Gastroenterol Nutr. 2020 May;70(5):664-680. doi: 10.1097/MPG.0000000000002655. PMID 32332478
- [Result] Alfaleh K, Anabrees J, Bassler D, Al-Kharfi T. Probiotics for prevention of necrotizing enterocolitis in preterm infants. Cochrane Database Syst Rev. 2011 Mar 16;(3):CD005496. doi: 10.1002/14651858.CD005496.pub3. PMID 21412889
- [Result] Wood NS, Marlow N, Costeloe K, Gibson AT, Wilkinson AR. Neurologic and developmental disability after extremely preterm birth. EPICure Study Group. N Engl J Med. 2000 Aug 10;343(6):378-84. doi: 10.1056/NEJM200008103430601. PMID 10933736
- [Result] Hortensius LM, van Elburg RM, Nijboer CH, Benders MJNL, de Theije CGM. Postnatal Nutrition to Improve Brain Development in the Preterm Infant: A Systematic Review From Bench to Bedside. Front Physiol. 2019 Jul 26;10:961. doi: 10.3389/fphys.2019.00961. eCollection 2019. PMID 31404162
- [Result] Cryan JF, O'Mahony SM. The microbiome-gut-brain axis: from bowel to behavior. Neurogastroenterol Motil. 2011 Mar;23(3):187-92. doi: 10.1111/j.1365-2982.2010.01664.x. PMID 21303428
- [Result] Yang I, Corwin EJ, Brennan PA, Jordan S, Murphy JR, Dunlop A. The Infant Microbiome: Implications for Infant Health and Neurocognitive Development. Nurs Res. 2016 Jan-Feb;65(1):76-88. doi: 10.1097/NNR.0000000000000133. PMID 26657483
- [Result] Huang EJ, Reichardt LF. Neurotrophins: roles in neuronal development and function. Annu Rev Neurosci. 2001;24:677-736. doi: 10.1146/annurev.neuro.24.1.677. PMID 11520916
- [Result] Ranuh R, Athiyyah AF, Darma A, Risky VP, Riawan W, Surono IS, Sudarmo SM. Effect of the probiotic Lactobacillus plantarum IS-10506 on BDNF and 5HT stimulation: role of intestinal microbiota on the gut-brain axis. Iran J Microbiol. 2019 Apr;11(2):145-150. PMID 31341569
- [Result] Nikolaou KE, Malamitsi-Puchner A, Boutsikou T, Economou E, Boutsikou M, Puchner KP, Baka S, Hassiakos D. The varying patterns of neurotrophin changes in the perinatal period. Ann N Y Acad Sci. 2006 Dec;1092:426-33. doi: 10.1196/annals.1365.041. PMID 17308169
- [Result] Liu DY, Shen XM, Yuan FF, Guo OY, Zhong Y, Chen JG, Zhu LQ, Wu J. The Physiology of BDNF and Its Relationship with ADHD. Mol Neurobiol. 2015 Dec;52(3):1467-1476. doi: 10.1007/s12035-014-8956-6. Epub 2014 Oct 30. PMID 25354496
- [Result] Jacobs SE, Hickey L, Donath S, Opie GF, Anderson PJ, Garland SM, Cheong JLY; ProPremsStudy Groups. Probiotics, prematurity and neurodevelopment: follow-up of a randomised trial. BMJ Paediatr Open. 2017 Nov 25;1(1):e000176. doi: 10.1136/bmjpo-2017-000176. eCollection 2017. PMID 29637171
- [Result] Chou IC, Kuo HT, Chang JS, Wu SF, Chiu HY, Su BH, Lin HC. Lack of effects of oral probiotics on growth and neurodevelopmental outcomes in preterm very low birth weight infants. J Pediatr. 2010 Mar;156(3):393-6. doi: 10.1016/j.jpeds.2009.09.051. Epub 2009 Nov 14. PMID 19914635
- [Result] Romeo MG, Romeo DM, Trovato L, Oliveri S, Palermo F, Cota F, Betta P. Role of probiotics in the prevention of the enteric colonization by Candida in preterm newborns: incidence of late-onset sepsis and neurological outcome. J Perinatol. 2011 Jan;31(1):63-9. doi: 10.1038/jp.2010.57. Epub 2010 Apr 22. PMID 20410904
- [Result] Sari FN, Eras Z, Dizdar EA, Erdeve O, Oguz SS, Uras N, Dilmen U. Do oral probiotics affect growth and neurodevelopmental outcomes in very low-birth-weight preterm infants? Am J Perinatol. 2012 Sep;29(8):579-86. doi: 10.1055/s-0032-1311981. Epub 2012 May 7. PMID 22566113
- [Result] Johnson S, Hollis C, Kochhar P, Hennessy E, Wolke D, Marlow N. Psychiatric disorders in extremely preterm children: longitudinal finding at age 11 years in the EPICure study. J Am Acad Child Adolesc Psychiatry. 2010 May;49(5):453-63.e1. PMID 20431465

DOCUMENTS (2):
  • Study Protocol (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT05945017/Prot_000.pdf
  • Informed Consent Form (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT05945017/ICF_001.pdf